CLINICAL TRIAL: NCT07151729
Title: Use of Anodal Transcranial Direct Current Stimulation to Enhance Upper Limb Recovery in Stroke
Brief Title: Use of Anodal tDCS to Enhance Upper Limb Recovery in Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Ng Teng Fong Healthcare Innovation Programme (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DSRB 2024-4011
Record Dates: First submitted 2025-08-08; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-05

CONDITIONS: Stroke
Keywords: stroke; tdcs; upper limb
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
  1 control group (with sham transcranial direct current stimulation) and 1 intervention group (with real anodal transcranial direct current stimulation)
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Anodal tDCS (Experimental): Anodal tDCS to contralateral dorsal premotor cortex (dPMc)
  Interventions: Device: Anodal tDCS
- Sham tDCS (Sham Comparator): Sham tDCS to contralateral dorsal premotor cortex (dPMc)
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Anodal tDCS — This anodal tDCS is applied over the contralateral dorsal premotor cortex (instead of the ipsilateral motor cortex in previous studies).
  Other Names: tDCS
  Arms: Anodal tDCS
Device: Sham tDCS — Sham tDCS is applied
  Other Names: tdcs
  Arms: Sham tDCS

SUMMARY:
This will be a randomized, blinded, sham-controlled trial. The medical device used, Soterix Medical 1x1 tDCS stimulator, is capable of delivering either real or sham tDCS and has been used in many randomised controlled trials in stroke patients.

50 patients with subacute stroke and severe upper limb weakness within 8 weeks of stroke on transfer to TTSH stroke rehab wards will be recruited over a period of 10 months. Recruited patients will be randomized into the intervention and control arms in a 1:1 ratio.

DETAILED DESCRIPTION:
The primary objective is to determine the clinical efficacy, technical feasibility and safety of anodal tDCS therapy to the unaffected hemisphere in hospitalized subacute stroke patients with severe arm weakness.

ELIGIBILITY:
Inclusion Criteria:

* First ever unilateral ischaemic or haemorrhagic stroke, as documented by CT or MRI scans
* Age 21-80 years, both males and females
* Within 8 weeks of stroke onset
* Severe weakness of one upper limb, defined by a Shoulder Abduction and Finger Extension (SAFE) score < 5 (Medical Research Council grading)
* Provision of informed consent by patient or a legal guardian in accordance with the local ethics committee guidelines and the Declaration of Helsinki

Exclusion Criteria:

* Bilateral hemispheric or cerebellar strokes
* Pre-existing arm pathology (e.g. contracture, severe pain, etc.) on the affected side
* Presence of brain implants, and previous insertion of external ventricular drains.
* Metallic implants at the level of the neck, mouth cavity and below are permitted (e.g. Cardiac stents, dental implants, pacemakers and other metallic objects)
* A history of spontaneous seizures, epilepsy, brain tumour, and cranial surgery
* Severe cognitive impairment (MOCA Score <10) that would hinder sufficient understanding of the instructions
* Pregnancy

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Upper Limb | At baseline (Day 0) At end of 10 tDCS sessions (Day 10) At 3 months after the 10th tDCS session (Month 3)
  Fugl-Meyer Upper Limb

SECONDARY OUTCOMES:
Streamlined Wolf Motor Function Test (sWMFT) | At baseline (Day 0) At end of 10 tDCS sessions (Day 10) At 3 months after the 10th tDCS session (Month 3)
  Streamlined Wolf Motor Function Test (sWMFT)
Functional Independence Measure (FIM) | At baseline (Day 0) At end of 10 tDCS sessions (Day 10)
  Functional Independence Measure (FIM) is a widely used objective assessment tool in rehabilitation to evaluate a patient's functional abilities and track their progress. It is a 18-item, 7-level scale, with higher scores indicating greater independence. The total FIM score ranges from 18 to 126.
EQ5D-5L | At baseline (Day 0) and at 3 months after the 10th tDCS session (Month 3)
  The EurolQol 5-Dimension 5-Level (EQ5D-5L) is a widely-used, non-disease specific questionnaire designed to assess a patient's health related quality of life. It serves as a patient-reported outcome instrument, capturing the patient's own perspective on their health. It consists of a descriptive system of five questions (each scored from Level 1 to 5, with a higher score indicating more severe problems) and a visual analogue scale (VAS) for overall health assessment. A higher VAS (from 0 to 100) would indicate a better quality of life.
Rate of Adverse Events from tDCS | Immediately after each tDCS session (total 10 sessions of tDCS)
  An adverse events questionnaire is administered immediately after each tDCS session. As such, each participant would fill up 10 adverse effects questionnaires after a total of 10 tDCS sessions.
  The rate of adverse events from tDCS would be computed from the number of adverse events divided by the total number of tDCS sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Tan Tock Seng Hospital - Integrated Care Hub, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
To protect the privacy of participants. Preparing IPD for sharing can also be time-consuming and resource-intensive.